CLINICAL TRIAL: NCT00464087
Title: Switching From Arixtra (Fondaparinux) to Angiomax (Bivalirudin) or Unfractionated Heparin in Patients With Acute Coronary Syndromes (ACS) Without ST-segment Elevation Undergoing Percutaneous Coronary Intervention (PCI): SWITCH III
Brief Title: Switching From Fondaparinux to Bivalirudin or Unfractionated Heparin in ACS Patients Undergoing PCI
Acronym: SWITCHIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWITCH III
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin (Active Comparator): Patients are switched from fondaparinux to heparin, receiving a dose of 60 U/Kg IV during the PCI
  Interventions: Drug: Switching from Fondaparinux to Bivalirudin or Unfractionated Heparin
- Bivalirudin (Active Comparator): Patients switched from fondaparinux to bivalirudin, received a bolus of 0.75 mg/kg IV followed by infusion of 1.75 mg/g per hour infusion during the PCI.
  Interventions: Drug: Switching from Fondaparinux to Bivalirudin or Unfractionated Heparin

INTERVENTIONS:
Drug: Switching from Fondaparinux to Bivalirudin or Unfractionated Heparin

SUMMARY:
The primary objective of this clinical trial is to evaluate safety of switching from fondaparinux to either unfractionated heparin or bivalirudin for patients experiencing acute coronary syndrome undergoing percutaneous coronary angioplasty.

DETAILED DESCRIPTION:
This is a prospective open label, randomized, multi-center registry. One hundred patients who received fondaparinux within the 24 hours prior to presentation to the coronary catheterization lab and who are suitable for percutaneous coronary intervention. The patients will be randomized in a 1:1 fashion to either unfractionated heparin or bivalirudin during the angioplasty. All patients will be followed throughout the duration of the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is, male or female, > 18 years of age; 2. The patient presents with coronary syndrome, unstable angina or non ST segment elevated myocardial infarction (NSTEMI) defined as at least one of the following criteria:

* Elevated creatine kinase MB or Troponin I or T (above ULN)
* ECG changes indicative of ischemia 3. The patient is scheduled for angiography, with possible angioplasty, evaluation of their coronary disease; 4. The patient is able and willing to conform to the requirements of the study and voluntarily signs an Informed Consent.

  1. ST elevated myocardial infarction within the preceding 48 hours;
  2. Patient weighs more than 400 lbs (181.2 kg) or less than 110 lbs (50 kg);
  3. Patients presenting on or received bivalirudin, GP IIb/IIIa inhibitors or low-molecular weight heparin within the preceding 24 hours;
  4. Patients that received unfractionated heparin less than or equal to 90 minutes prior to fondaparinux administration.
  5. Patients with known conditions of bleeding diathesis or actively bleeding within the previous 6 months (GI bleed etc.);
  6. Known diagnosis of acute bacterial endocarditis;
  7. Patients with cardiogenic shock or required intra-aortic balloon pump (IABP)
  8. If patient is on warfarin (Coumadin) therapy;
  9. Patients who had a major or minor stroke (CVA or TIA) or major surgery within the past 6 months;
  10. Known impaired renal function (creatinine ≥ 3.0 mg/dL (265.2 μmol/L),) status post renal transplant, patients on chronic dialysis or creatinine clearance ≤ 30 ml/min;
  11. A platelet count of less than 100,000 cells/mm3;
  12. Known allergies to fondaparinux, aspirin, clopidogrel bisulfate (PlavixR), ticlopidine (TiclidR), heparin, bivalirudin, or contrast that cannot be medically managed;
  13. Prior angioplasty within the previous 30 days;
  14. Contraindication to low-molecular weight heparin, unfractionated heparin or bivalirudin;
  15. Pregnant or lactating women;
  16. Any significant medical condition, which in the investigator's opinion, may interfere with the patient's optimal participation in the study;
  17. Currently participating in an investigational drug or another device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Washington Hospital Center, Washington, DC
Locations (7):
- United States (5):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Institut Universitaire de cardiologie et de Pneumologie de Québec (Hôpital Laval), Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who were enrolled and received fondaparinux and who did not have sufficient disease requiring any revascularization procedure will be followed through the duration of the hospitalization. Patients will have a complete blood count (CBC) prior to discharge. These patients are enrolled, but considered screen failures.
Groups:
- Heparin: All patients received fondaparinux at a dose of 2.5 mg subcutaneously no more than 24 hours before angioplasty. They are randomized to unfractionated heparin during angioplasty and receive a minimum dose of 60 U/kg IV.
- Bivalirudin: All patients received fondaparinux at a dose of 2.5 mg subcutaneously no more than 24 hours before angioplasty. They are randomized to Bivalirudin during angioplasty and receive a minimum dose of bolus 0.75 mg/kg IV followed by, infusion of 1.75 mg/kg/hr for the duration of the PCI.
- Screen Failures: These patients were enrolled because they received study drug, but did not have enough disease to require PCI.
Period: Overall Study
Arm/Group | Heparin | Bivalirudin | Screen Failures
Started | 49 | 51 | 29
Completed | 49 | 51 | 0
Not Completed | 0 | 0 | 29
Not completed — No PCI per inclusion criteria | 0 | 0 | 29

BASELINE CHARACTERISTICS:
Groups:
- Heparin: unfrationated heparin during angioplasty
- Bivalirudin: bivalirudin during angioplasty
- Screen Failures: Screen Failures are patients who are enrolled and receive the study drug, but do not have enough disease to have percutaneous coronary intervention.
- Total: Total of all reporting groups
Arm/Group | Heparin | Bivalirudin | Screen Failures | Total
Number analyzed (Participants) | 49 | 51 | 29 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 27 | 22 | 80
  >=65 years | 18 | 24 | 7 | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 62.18 (13.36) | 63.33 (12.17) | 54.45 (13.62) | 60.45 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 8 | 40
  Male | 31 | 37 | 21 | 89
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 29 | 63
  Canada | 33 | 33 | 0 | 66

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be in Hospital Major Bleed as Defined by the Study Protocol, Assessed at Three Time Points: After Study Drug Administration, But Prior to Randomization;After Randomization During PCI; and After PCI, Prior to Discharge
Description: Characterized as Fatal bleed, Major bleed (SWITCH III criteria) or major bleed (OASIS criteria)
Time Frame: During hospitalization, after Fondaparinux administration, prior to randomization
Measure: Number; unit: participants
Groups:
- Heparin: unfractionated heparin during angioplasty
Arm/Group | Heparin | Bivalirudin | Screen Failures
Number analyzed (Participants) | 49 | 51 | 0
participants | 0 | 0 |

2. Secondary Outcome: Secondary in Hospital Endpoint Will be In-hospital Death (Non-hemorrhagic Related), Vascular Access Site Complications, Myocardial Infarction, Need for Repeat Revascularization, Procedural Complication and Catheter Thrombosis
Description: Characterized as death, access site complication, access site thrombus, hematoma, myocardial infarction, repeat vascularization, dissection, stent thrombosis, catheter thrombosis
Time Frame: during index hospitalization
Measure: Number; unit: participants
Arm/Group | Heparin | Bivalirudin
Number analyzed (Participants) | 49 | 51
participants | 4 | 4

3. Primary Outcome: The Primary Endpoint Will be in Hospital Major Bleed as Defined by the Study Protocol, Assessed at Three Time Points: After Study Drug Administration, But Prior to Randomization;After Randomization During PCI; and After PCI, Prior to Discharge
Description: Categorized as Fatal bleed, major bleed (SWITCH III criteria) or major bleed (OASIS criteria)
Time Frame: During hospitalization, after randomization, during PCI
Measure: Number; unit: participants
Arm/Group | Heparin | Bivalirudin | Screen Failures
Number analyzed (Participants) | 49 | 51 | 0
participants | 0 | 0 |

4. Primary Outcome: The Primary Endpoint Will be in Hospital Major Bleed as Defined by the Study Protocol, Assessed at Three Time Points: After Study Drug Administration, But Prior to Randomization;After Randomization During PCI; and After PCI, Prior to Discharge
Description: Characterized as fatal bleed, major bleed (SWITCH III criteria) or major bleed (OASIS criteria)
Time Frame: During hospitalization, after PCI
Measure: Number; unit: participants
Arm/Group | Heparin | Bivalirudin | Screen Failures
Number analyzed (Participants) | 49 | 51 | 0
participants | 0 | 1 |

ADVERSE EVENTS:
Arm/Group | Heparin | Bivalirudin | Screen Failures
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/51 | 0/0
Other Adverse Events (participants affected / at risk) | 4/49 | 4/51 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin (N=49) | Bivalirudin (N=51) | Screen Failures (N=0)
Major Bleed (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin (N=49) | Bivalirudin (N=51) | Screen Failures (N=0)
Access Site Complication (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Dissection (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Repeat revascularization (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial included only small number of patients and is not powered to detect intergroup differences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No